CLINICAL TRIAL: NCT01318954
Title: The Effect of Allergen Immunotherapy on Exhaled Nitric Oxide in Adult Patients With Asthma and Allergic Rhinitis
Status: Completed | Type: Observational
Sponsor: Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C. (Other)
Responsible Party: Principal Investigator, Michele Columbo, M.D., Principal Investigator, Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Other Study IDs: F/N-R07-2592B
Record Dates: First submitted 2009-09-28; First posted 2011-03-21 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Allergic Asthma; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Desensitization, Immunologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects on allergen immunotherapy: Measurements of Nitric Oxide by NIOX MINO. This device is now FDA approved.
  Interventions: Biological: Allergen immunotherapy

INTERVENTIONS:
Biological: Allergen immunotherapy

SUMMARY:
This study will evaluate whether exhaled nitric oxide levels are affected by allergen immunotherapy ("allergy shots"). The investigators' hypothesis is that successful allergen immunotherapy may be accompanied by decreased exhaled nitric oxide levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years old with allergic asthma and/or allergic rhinitis who are beginning allergen desensitization

Exclusion Criteria:

* Smokers
* Subjects of dimished capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with allergic asthma and allergic rhinitis undergoing allergen immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of allergen immunotherapy on exhaled nitric oxide | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michele Columbo, M.D., Principal Investigator — Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Locations (1):
- Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C., Bryn Mawr, Pennsylvania, United States